CLINICAL TRIAL: NCT03704012
Title: Assessment of the Efficacy of Massage and Kinesiotherapy Applied by the Parents on the Biological State, Neuromotor Activity and Other Associated Factors in Hospitalized Premature Birth (PreMas)
Brief Title: Efficacy of Massage Applied by the Parents in Hospitalized Premature Birth (PreMas)
Acronym: PreMas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, María José Álvarez Álvarez, Collaborating Professor, Nursing and Physical Therapy Department, Universidad de León (Spain), Universidad de León
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PI12/02763
Record Dates: First submitted 2018-02-23; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Massage; Premature Infant; Premature Birth; Preterm Infant
Keywords: Premature Infant; Massage; Tactile Kinesthetic Stimulation
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Intervention Model Description: The control group included all preterm infants from months 1-6 and 19-24 of the study. The intervention group included all the premature newborns from the 7-18 months of the study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (No Intervention): Control Group receives routine care.
- Massage and kinesiotherapy (Experimental): Intervention Group, receives massage and kinesiotherapy. Behavioral: Protocol of massage therapy and kinesiotherapy. Infants received massage and kinesiotherapy twice a day; 15 minutes each.
  Interventions: Behavioral: Protocol of massage therapy and kinesiotherapy

INTERVENTIONS:
Behavioral: Protocol of massage therapy and kinesiotherapy — Infants received massage and kinesiotherapy, applied by parents, twice a day; 15 minutes each.
  Other Names: Massage; Massage Therapy; Tactile Kinesthetic Stimulation
  Arms: Massage and kinesiotherapy

SUMMARY:
The purpose of this study was to analyze the efficacy of massage therapy and kinesiotherapy, applied by the parents of hospitalized preterm infants, in the improvement of the biological state, neuromotor activity and other associated factors.

DETAILED DESCRIPTION:
Premature infants are prematurely deprived of the cutaneous stimulation provided during intrauterine development and of the continuous contact with their parents. It has and adverse effect on both psychological and biological development of the child.

Knowledge of these factors has led many neonatal units to begin to introduce therapeutic massage protocols to facilitating satisfactory neuromotor and anthropometric development of preterm infants.

In this study, premature newborns were assigned to one of two groups:

A: Control Group. B: Massage and kinesiotherapy Group, 15 minutes twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 26 to 37 gestational weeks.
* Low birth weight, less than 2249 grams.
* Weight of at least 1250 grams at time of entry into study.
* Must be at least 48 hours of age.
* Must have hemodynamic stability.
* Absence of congenital and genetic anomalies.
* Absence of alterations of the central nervous system.
* Intact skin.
* Stable parameters (according to the neonatologist´s criteria) to participate in the intervention.

Exclusion Criteria:

* Family refusal to participate in the study.
* High frequency mechanical ventilation.
* Fraction of Inspired Oxygen (FiO2)>70%.
* Inotropic support.
* Septic shock.
* Persistent tachycardia.
* Persistent bradycardia.
* Gastrointestinal disorders.

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-01-02 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Effect on weight | From baseline to hospital discharge, approximately 10 days
  Effect of treatment on weight
Effect of lenght | From baseline to hospital discharge, approximately 10 days
  Effect of treatment on lenght
Effect on head circumference | From baseline to hospital discharge, approimately 10 days
  Effect of treatment on head circumference
Effect on neuromotor development | From baseline to up to 37 gestational weeks
  Effect of treatment on neuromotor development. Neuromotor development were measured using the Spanish Premie-Neuro Scale, a scale for the neurological examination of premature babies, between 23 and 37 gestational weeks.
  It consists of twenty-four items divided into three factors: Neurological, movement and responsiveness, each with eight items. Each of the items is assigned a score of 1, 3 or 5. The scores for items are added up to yield a total raw score, with the possible figures for this ranging from 24 to 120 (higher values represent a better neuromotor development).

SECONDARY OUTCOMES:
Average daily weight gain | From baseline to hospital discharge, approimately 10 days
  Effect of treatment on daily weight gain during the hospitalization period

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fernández-García, PhD, Principal Investigator — Proffesor. Nursing and Physical Therapy Department. University of León.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alvarez MJ, Fernandez D, Gomez-Salgado J, Rodriguez-Gonzalez D, Roson M, Lapena S. The effects of massage therapy in hospitalized preterm neonates: A systematic review. Int J Nurs Stud. 2017 Apr;69:119-136. doi: 10.1016/j.ijnurstu.2017.02.009. Epub 2017 Feb 14. PMID 28235686
- [Result] Fernandez D, Alvarez MJ, Rodriguez D, Rodriguez M, Fernandez E, Urdiales P. Spanish Validation of the Premie-Neuro Scale in Premature Infants. J Pediatr Nurs. 2015 Jul-Aug;30(4):560-7. doi: 10.1016/j.pedn.2014.11.002. Epub 2014 Nov 26. PMID 25433214
- [Derived] Alvarez-Alvarez MJ, Fernandez-Garcia D, Gomez-Salgado J, Ordas B, Rodriguez-Gonzalez MD, Martinez-Isasi S. Effectiveness of the application of massage therapy and kinesitherapy by parents on premature neonates: A research protocol. J Adv Nurs. 2019 Nov;75(11):3097-3104. doi: 10.1111/jan.14135. Epub 2019 Jul 30. PMID 31236954